CLINICAL TRIAL: NCT06156943
Title: Advanced Goal-Directed Impedancemetry Strategy for Lung Resection Surgery : a Multicenter, Randomized, Controlled Trial (AEGIS Study)
Brief Title: Advanced Goal-Directed Impedancemetry Strategy for Lung Resection Surgery
Acronym: AEGIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 69HCL22_1133; 2024-A01843-44 (Other: ID-RCB)
Record Dates: First submitted 2023-11-20; First posted 2023-12-05 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: High-risk Lung Resection Surgery
Keywords: goal-directed fluid therapy; Chest bioreactance; lung resection surgery

STUDY DESIGN:
Intervention Model Description: National prospective multicenter randomized simple blind controlled study comparing a standard of care (control group) to an individualized strategy of intraoperative GDFT driven by non-invasive continuous SV monitoring via chest bioreactance (optimized group).
Who Masked: Participant
Masking Description: The patients are the only ones masked. As double blind is not possible, an adjudication committee, whose members will be unaware of the procedure assignments, will adjudicate all the clinical outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Optimized group managed by the Starling device (Experimental): In the optimized group, patients will be managed intraoperatively with the Starling device according to the Société Française d'Anesthésie Réanimation 2024 GDFT protocol (Alter C. https://sfar.org/optimisation-hemodynamique-perioperatoire-adulte-dont-obstetrique/). It is a non-invasive fluid management monitoring system provides continuous hemodynamic monitoring and empowers fluid management across the continuum of care. Thanks to this device, patients will be managed according to the following protocol: fluid responsiveness will be systematically assessed after anesthetic induction and throughout the procedure as soon as the basal SV monitored by the Starling device decrease by at least 10%. To do so, repetitive fluid challenges (200 ± 50 ml of cristalloids) will be quickly delivered until SV stops to increase by 10% or more. Vasoactive and/or inotropic agents will be used at the discretion of the attending anesthesiologists in case of fluid unresponsiveness.
  Interventions: Procedure: individualized goal-directed fluid therapy by Starling device
- Control group managed by standard of care (Other): In the control group, patients will be managed intraoperatively at the discretion of the attending anesthesiologists, in accordance with their institutional protocols (i.e. fluids and/or vasoactive agents are given to maintain mean arterial pressure ≥ 65 mmHg).
  Interventions: Procedure: group managed by standard of care

INTERVENTIONS:
Procedure: individualized goal-directed fluid therapy by Starling device — For patients in optimized group, fluids will be managed by Starling device during the lung resection surgery.
  Arms: Optimized group managed by the Starling device
Procedure: group managed by standard of care — Patients will be managed intraoperatively at the discretion of the attending anesthesiologists, in accordance with their institutional protocols
  Arms: Control group managed by standard of care

SUMMARY:
High-risk patients scheduled for lung resection surgery are increasing and theoretically eligible to perioperative individualized goal-directed fluid therapy (GDFT). However, thoracic surgery is challenging for intraoperative stroke volume (SV) and/or cardiac output monitoring because it requires lateral positioning, one-lung ventilation, and open-chest condition. Pulse contour analysis and esophageal Doppler have been proposed with contrasting results, whereas dynamic indices have been shown useless for predicting fluid responsiveness in that specific setting. Besides, more invasive technologies like thermodilution are not routinely used at the bedside by careproviders.

Chest bioreactance seems to be a feasible, safe, rustic, easy-to-use, and plug-and-play method to non-invasively and continuously monitor SV and cardiac output in thoracic cancer surgery patients, able to detect significant spontaneous and pharmacologically-induced changes over time. The impact of chest bioreactance on patients 'outcome remains however to be demonstrated.

Indeed, the routine fluid management in patients undergoing lung resection surgery could be responsible of hypovolemia/hypoperfusion and/or hypervolemia/congestion leading to postoperative complications.

The present national prospective multicenter randomized simple blind study aims to demonstrate that an individualized goal-directed fluid therapy (GDFT) driven by chest bioreactance improves outcomes within 30 days in lung resection surgery patients when compared with a standard of care. As double blind is not possible, an adjudication committee, whose members will be unaware of the procedure assignments, will adjudicate all the clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years old)
* High-risk patients (ASA score ≥ 3 and/or ventilatory deficit (defined as FEV1≤70% and/or VC≤70%) and/or AKI risk index ≥ III and/or modified clinical Lee Criteria ≥2) undergoing elective open-chest or video-assisted or robotic lung resection surgery
* Patients who have provided written informed consent to participate in the study
* Patients affiliated with a social health insurance

Exclusion Criteria:

* Pleural or mediastinal resection surgery
* Emergency surgery (Less than 24h)
* Patients unable to understand the purpose of the study
* Patients participating in another trial that would interfere with this study
* Female patients who are pregnant, lactating or women of child-bearing potential without effective methods of contraception
* Female patients with positive β-HCG blood test
* Patients under judicial protection (guardianship, curatorship)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 722 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
A composite of postoperative complications rate adapted from the Clavien-Dindo classification with only events ≥ class II | Within 30 days after the surgery
  It will be performed in each group and assessed by an independent adjudication committee.
  Clavien-Dindo classification :
  Class II :
  * Pulmonary complications (any infection requiring antibiotics, non-invasive ventilation)
  * Cardiovascular complications (postoperative atrial fibrillation (POAF) requiring treatment, deep venous thrombosis)
  * Renal complications (acute kidney injury (AKI), defined as an increase of serum creatinine of more than 50% or more than 26.5 µmol/L, requiring fluid supply or diuretics)
  * Cerebral complications (delirium requiring treatment, stroke)
  * Blood products transfusion Class III
  * Reoperation from any cause Class IV
  * Any unscheduled admission to the intensive care unit (ICU) Class V
  * Mortality from any cause The analysis of the main endpoint will be performed by a mixed logistic regression model. It will take into account as explanatory variable the intervention, as well as the type of surgery (open-chest or video-assisted or robotic). It will include

SECONDARY OUTCOMES:
Each item of the primary composite endpoint between both groups | Within 30 days after the surgery
  Items of the primary composite endpoint :
  - Pulmonary complications rate
  Each item of the primary composite endpoint will be described in each group in terms of number/percentage of patients and compared using the chi-2 test or the exact test of Fisher. An Holm correction will be applied to take into account multiple testing.
Each item of the primary composite endpoint between both groups | Within 30 days after the surgery
  Items of the primary composite endpoint :
  - Cardiovascular complications rate
  Each item of the primary composite endpoint will be described in each group in terms of number/percentage of patients and compared using the chi-2 test or the exact test of Fisher. An Holm correction will be applied to take into account multiple testing.
Each item of the primary composite endpoint between both groups | Within 30 days after the surgery
  Items of the primary composite endpoint :
  - Renal complications rate
  Each item of the primary composite endpoint will be described in each group in terms of number/percentage of patients and compared using the chi-2 test or the exact test of Fisher. An Holm correction will be applied to take into account multiple testing.
Each item of the primary composite endpoint between both groups | Within 30 days after the surgery
  Items of the primary composite endpoint :
  - Cerebral complications rate
  Each item of the primary composite endpoint will be described in each group in terms of number/percentage of patients and compared using the chi-2 test or the exact test of Fisher. An Holm correction will be applied to take into account multiple testing.
Each item of the primary composite endpoint between both groups | Within 30 days after the surgery
  Items of the primary composite endpoint :
  - Blood products transfusion rate
  Each item of the primary composite endpoint will be described in each group in terms of number/percentage of patients and compared using the chi-2 test or the exact test of Fisher. An Holm correction will be applied to take into account multiple testing.
Each item of the primary composite endpoint between both groups | Within 30 days after the surgery
  Items of the primary composite endpoint :
  - Reoperation from any cause rate
  Each item of the primary composite endpoint will be described in each group in terms of number/percentage of patients and compared using the chi-2 test or the exact test of Fisher. An Holm correction will be applied to take into account multiple testing.
Each item of the primary composite endpoint between both groups | Within 30 days after the surgery
  Items of the primary composite endpoint :
  - Any admission to the ICU rate
  Each item of the primary composite endpoint will be described in each group in terms of number/percentage of patients and compared using the chi-2 test or the exact test of Fisher. An Holm correction will be applied to take into account multiple testing.
Each item of the primary composite endpoint between both groups | Within 30 days after the surgery
  Items of the primary composite endpoint :
  - Mortality rate
  Each item of the primary composite endpoint will be described in each group in terms of number/percentage of patients and compared using the chi-2 test or the exact test of Fisher. An Holm correction will be applied to take into account multiple testing.
Length of stay in hospital (days) and number/percentage of patients with length of stay in hospital ≥ 5 days in each group | 5 days
  Quantitative secondary endpoints will be described in each group, and will be compared between the two groups using the t test of Student or the test of Mann and Whitney, according to the shape of the distribution.
  Qualitative secondary outcome will be described in each group by the number/percentage of patients and compared using the chi-2 test or the exact test of Fisher.
APGAR surgical score and number/percentage of patients with APGAR surgical score < 7 in each group | 1 day
  Quantitative secondary endpoints will be described in each group, and will be compared between the two groups using the t test of Student or the test of Mann and Whitney, according to the shape of the distribution.
  Qualitative secondary outcome will be described in each group by the number/percentage of patients and compared using the chi-2 test or the exact test of Fisher.

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Hopital Louis Pradel, Bron
  - CHU Dijon Bourgogne, Dijon
  - Hôpital Arnaud de Villeneuve - CHU Montpellier, Montpellier
  - Chu Nancy, Nancy
  - Hôpital Européen Georges Pompidou, Paris
  - Hopital du Haut-Leveque - CHU Bordeaux, Pessac
  - CHU de Rennes, Rennes
  - CHU Nantes, Saint-Herblain
  - CHU Strasbourg, Strasbourg
  - Chu Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No